CLINICAL TRIAL: NCT02468648
Title: Investigation of Viral Kinetics, Interferon Stimulated Genes (ISGs) and mirRNA Among Subjects Infected With Different Hepatitis C Virus Genotypes During Therapy With Sofosbuvir and GS-5816
Brief Title: Viral Kinetics, Interferon Stimulated Genes (ISGs) and mirRNA Among Subjects Infected With Different Hepatitis C Virus Genotypes During Therapy With Sofosbuvir and GS-5816
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: National Institute of Diabetes and Digestive and Kidney Diseases (NIDDK) (NIH)
Responsible Party: Sponsor
Organization: National Institutes of Health Clinical Center (CC) (NIH)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 150143; 15-DK-0143
Record Dates: First submitted 2015-06-09; First posted 2015-06-11 (Estimated); Results first posted 2020-03-19 (Actual); Last update posted 2020-03-19 (Actual); Status verified 2018-09-14

CONDITIONS: Chronic Hepatitis C
Keywords: Oral Therapy; Liver Biopsy; Chronic Hepatitis C
MeSH Terms: conditions — Hepatitis C, Chronic | interventions — Sofosbuvir; velpatasvir

STUDY DESIGN:
Oversight: FDA-regulated Drug: Yes

ARMS (1):
- Combination of sofosbuvir and GS-5816 (Experimental): Combination of sofosbuvir and GS-5816 agent into a single pill will be used.
  Interventions: Drug: Sofosbuvir; Drug: GS-5816

INTERVENTIONS:
Drug: Sofosbuvir — An NS5B polymerase inhibitor that is already approved for use in combination with interferon and ribavirin for the treatment of HCV genotype 1 infection
Drug: GS-5816 — An NS5A replication complex inhibitor with potent activity against most strains of hepatitis C virus.

SUMMARY:
Background:

- Chronic hepatitis C is a serious liver disease. Current treatments have side effects. New drugs have been developed, but they work better in some people than others. Researchers want to learn why.

Objective:

- To learn why new hepatitis C drugs sometimes do not work. Also, to learn if these drugs are safe and how well they work in people with different virus strains.

Eligibility:

- Adults age 18 and older who are infected with hepatitis C virus genotypes 1-4 and who have either never been treated or treated previously with an interferon regimen (with or without ribavirin) that failed to clear the virus.

Design:

* Participants will be screened with medical history and physical exam. They will have blood and urine tests and complete questionnaires.
* Participants will have a Fibroscan, an ultrasound that measures liver stiffness and other liver scans. They will have an electrocardiogram.
* Eligible participants will have a liver biopsy.
* Participants will be admitted to the Clinical Center. They will have a physical exam and blood tests, and complete questionnaires.
* They will take the first study drug dose as a tablet taken once daily.
* Participants will take the drug at home for 12 weeks.
* Participants will have 6 study visits. They will have blood and vital signs taken, and complete questionnaires.
* At week 4, participants will have another liver biopsy.
* After their last drug dose, participants will have 5 follow-up visits. They will have blood and vital signs taken, and complete questionnaires. They will discuss their medications and side effects. They may have another Fibroscan.

DETAILED DESCRIPTION:
Up to 140 patients with chronic hepatitis C, genotypes 1-4, who were never treated or previously treated but failed a course of therapy with any interferon and ribavirin combination regimen will be eligible to be enrolled into this pilot study to evaluate the combination of sofosbuvir and GS-5816 as a fixed dose tablet to improve response to antiviral therapy. To enrich the study population with subjects with a greater likelihood of virological relapse after stopping therapy, we plan to enroll a minimum of 60% treatment-experienced subjects and 50% with cirrhosis. These two drugs inhibit key enzymes that are necessary for viral replication. Sofosbuvir, an NS5B polymerase inhibitor is already approved for use in combination with interferon and ribavirin for the treatment of HCV genotype 1 infection. GS-5816 is an NS5A replication complex inhibitor with potent activity against most strains of hepatitis C virus. Combining these two agents into a single pill should improve patient compliance and improve tolerability because interferon and ribavirin will not be part of the regimen. After medical evaluation and liver biopsy, patients will receive combination therapy with sofosbuvir and GS-5816 one pill a day for 12 weeks. The baseline liver biopsy is necessary to assess the amount of liver damage caused by the HCV and to measure expression of genes associated with clearance of HCV. Blood samples will be collected to monitor safety and response to therapy and for research purposes. HCV RNA levels will be monitored frequently for the initial 4 weeks and then at monthly intervals for the remaining 8 weeks of antiviral therapy. All subjects will undergo a second liver biopsy, 4 weeks after starting therapy. The second biopsy is being performed for research purposes so investigators can determine specifically which liver genes are associated with failure of therapy (and response to therapy). Subjects who refuse the second liver biopsy will continue to receive SOF/GS-5816 treatment for the planned 12 week duration Patients in whom serum HCV RNA is greater than or equal to lower limit of quantification (LLOQ) after 2 consecutive HCV RNA < LLOQ or who have a confirmed > 1 log10 increase from nadir will discontinue therapy (because continuing therapy is considered futile i.e. it is unlikely to work). The major endpoints will be changes in interferon stimulated gene and protein expression in the liver and changes in HCV RNA levels in liver and serum between baseline and 4 weeks and rates of sustained virologic response at post-treatment week 12. Secondary endpoints will be safety and sustained virologic response at post-treatment week 24 weeks.

ELIGIBILITY:
* INCLUSION CRITERIA:

Subjects must meet all of the following inclusion criteria to be eligible for participation in this study.

* Willing and able to provide written informed consent.
* Male or female, age greater than or equal to18 years.
* Body mass index (BMI) greater than or equal to 18 kg/m^2.
* HCV RNA greater than or equal to10^4 IU/mL at Screening
* HCV genotypes 1a, 1b, 2, 3 or 4 at screening
* Confirmation of chronic HCV infection documented by either:

  * A positive anti-HCV antibody test or positive HCV RNA or positive HCV genotyping test at least 6 months prior to the Baseline/Day 1 visit, or
  * A liver biopsy performed within 12 weeks prior to the Baseline/Day 1 visit with evidence of chronic HCV infection. A prior biopsy would be acceptable if performed with 12 weeks AND liver tissue stored in RNALater was available.
* Screening ECG without clinically significant abnormalities.
* Subjects must have the following laboratory parameters at screening:

  * ALT less than or equal to 10 times the upper limit of normal (ULN)
  * AST less than or equal to 10 times ULN
  * Direct bilirubin less than or equal to 1.5 ULN
  * Platelets > 70,000
  * HbA1c less than or equal to8.5%
  * eGFR greater than or equal to 60 mL /min, as calculated by the CKD-EPI equation.
  * Hemoglobin greater than or equal to 10g/dL.
  * Albumin greater than or equal to 3g/dL
  * INR less than or equal to 1.5 x ULN unless subject has known hemophilia or is stable on an anticoagulant regimen affecting INR.
* A female subject is eligible to enter the study if it is confirmed that she is:

  * Not pregnant or nursing
  * Of non-childbearing potential (i.e., women who have had a hysterectomy, have both ovaries removed or medically documented ovarian failure, or are postmenopausal women > 50 years of age with cessation (for greater than or equal to 12 months) of previously occurring menses),

OR

* Of childbearing potential (i.e., women who have not had a hysterectomy, have not had both ovaries removed, and have not had medically documented ovarian failure). Women less than or equal to 50 years of age with amenorrhea will be considered to be of childbearing potential. These women must have a negative serum pregnancy test at Screening and a negative urine pregnancy test on the Baseline/Day 1 visit prior to randomization. They must also agree to one of the following from 3 weeks prior to Baseline/Day 1 until 90 days after last dose of study drug:

  * Complete abstinence from intercourse. Periodic abstinence from intercourse (e.g., calendar, ovulation, symptothermal, post-ovulation methods) is not permitted.
  * Consistent and correct use of 1 of the following methods of birth control listed below in addition to a male partner who correctly uses a condom from the date of Screening until 90 days after last dose of study drug:

    * intrauterine device (IUD) with a failure rate of < 1% per year
    * female barrier method: cervical cap or diaphragm with spermicidal agent
    * tubal sterilization
    * vasectomy in male partner
    * hormone-containing contraceptive:

      * implants of levonorgestrel
      * injectable progesterone
      * oral contraceptives (either combined or progesterone only)
      * contraceptive vaginal ring
      * transdermal contraceptive patch

        * All male study participants must agree to consistently and correctly use a condom, while their female partner agrees to use 1 of the methods of birth control listed above, from the date of Screening until 90 days after last dose of study drug.
        * Male subjects must agree to refrain from sperm donation from 90 days after their last dose of study drug.
        * Subject must be of generally good health, with the exception of chronic HCV infection, as determined by the Investigator.
        * Subject must be able to comply with the dosing instructions for study drug administration and able to complete the study schedule of assessments, including all required post treatment visits.

EXCLUSION CRITERIA:

Subjects who meet any of the following exclusion criteria will not to be enrolled in this study.

* Current or prior history of any of the following:

  * Clinically-significant illness (other than HCV) or any other major medical disorder that may interfere with subject treatment, assessment or compliance with the protocol; subjects currently under evaluation for a potentially clinically-significant illness (other than HCV) are also excluded.
  * Gastrointestinal disorder or post-operative condition that could interfere with the absorption of the study drug.
  * Difficulty with blood collection and/or poor venous access for the purposes of phlebotomy.
  * Clinical hepatic decompensation (i.e., ascites, encephalopathy or variceal hemorrhage).
  * Solid organ transplantation.
  * Significant pulmonary disease, significant cardiac disease or porphyria.
  * Psychiatric hospitalization, suicide attempt, and/or a period of disability as a result of their psychiatric illness within the last 5 years. Subjects with psychiatric illness (without the prior mentioned conditions) that is well-controlled on a stable treatment regimen for at least 12 months prior to randomization or has not required medication in the last 12 months may be included.
  * Malignancy within 5 years prior to screening, with the exception of specific cancers that are entirely cured by surgical resection (basal cell skin cancer, etc). Subjects under evaluation for possible malignancy are not eligible.
  * Significant drug allergy (such as anaphylaxis or hepatotoxicity).
* Any prior treatment with a direct acting antiviral agent (protease inhibitors, NS5A inhibitors and NS5B polymerase inhibitors/non-nucleoside polymerase inhibitors.)
* Pregnant or nursing female or male with pregnant female partner.
* Chronic liver disease of a non HCV etiology (e.g., hemochromatosis, Wilson s disease, alfa 1 antitrypsin deficiency, cholangitis).
* Infection with hepatitis B virus (HBV) or human immunodeficiency virus (HIV).
* Clinically-relevant drug abuse within 12 months of screening. A positive drug screen will exclude subjects unless it can be explained by a prescribed medication; the diagnosis and prescription must be approved by the investigator.
* Use of any prohibited concomitant medications as described within 21 days of the Baseline/Day 1 visit; this washout period does not apply to PPIs, which can be taken up to 7 days before baseline Day 1.
* Use of antiviral medications within the last 30 days.
* Chronic use of systemically administered immunosuppressive agents (e.g., prednisone equivalent > 10 mg/day).
* Known hypersensitivity to GS-5816, SOF, or formulation excipients.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 72 (Actual)
Dates: Start 2015-06-09; Primary Completion 2018-09-14 (Actual); Study Completion 2018-09-14 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Marc G Ghany, M.D., Principal Investigator — National Institute of Diabetes and Digestive and Kidney Diseases (NIDDK)
Locations (1):
- National Institutes of Health Clinical Center, 9000 Rockville Pike, Bethesda, Maryland, United States

REFERENCES:
- See also: NIH Clinical Center Detailed Web Page — https://clinicalstudies.info.nih.gov/cgi/detail.cgi?B_2015-DK-0143.html

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Combination of Sofosbuvir and GS-5816
Started | 72
Completed | 71
Not Completed | 1
Not completed — Death | 1

BASELINE CHARACTERISTICS:
Arm/Group | Combination of Sofosbuvir and GS-5816
Number analyzed (Participants) | 72
Age, Continuous [Mean (Standard Deviation); unit: years] | 58.1 (10.2)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 36
  Male | 36
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 1
  Asian | 8
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 19
  White | 40
  More than one race | 2
  Unknown or Not Reported | 2

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With Sustained Virologic Response
Description: Absence of detectable virus 12 weeks after completion of antiviral therapy
Time Frame: 12 weeks
Measure: Count of Participants; unit: Participants
Arm/Group | Combination of Sofosbuvir and GS-5816
Number analyzed (Participants) | 71
Participants | 70

2. Primary Outcome: Number of Participants Who Maintained HCV RNA Levels in Liver and Serum Less Than Lower Limit of Quantification (LLOQ)
Time Frame: 4 weeks
Measure: Count of Participants; unit: Participants
Arm/Group | Combination of Sofosbuvir and GS-5816
Number analyzed (Participants) | 71
Participants | 55

3. Secondary Outcome: Number of Participants Who Sustained Virologic Response
Description: Absence of detectable virus 24 weeks after completion of antiviral therapy
Time Frame: 24 weeks
Measure: Count of Participants; unit: Participants
Arm/Group | Combination of Sofosbuvir and GS-5816
Number analyzed (Participants) | 71
Participants | 70

4. Secondary Outcome: Number of Participants Who Maintained HCV RNA Levels in Liver and Serum Less Than Lower Limit of Quantification (LLOQ)
Time Frame: 24 weeks
Measure: Count of Participants; unit: Participants
Arm/Group | Combination of Sofosbuvir and GS-5816
Number analyzed (Participants) | 71
Participants | 70

ADVERSE EVENTS:
Time Frame: 24 months
Arm/Group | Combination of Sofosbuvir and GS-5816
All-Cause Mortality (participants affected / at risk) | 1/72
Serious Adverse Events (participants affected / at risk) | 2/72
Other Adverse Events (participants affected / at risk) | 67/72
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Combination of Sofosbuvir and GS-5816 (N=72)
Pain after a radiological biopsy and direct cannulation of the portal vein (Surgical and medical procedures) | 1 (1)
Small bowel obstruction (Gastrointestinal disorders) | 1 (1)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Combination of Sofosbuvir and GS-5816 (N=72)
Fatigue (General disorders) | 44 (204)
Headache (Nervous system disorders) | 47 (171)
Trouble sleeping (Nervous system disorders) | 36 (159)
Muscle pain (Musculoskeletal and connective tissue disorders) | 36 (142)
Iching (Skin and subcutaneous tissue disorders) | 31 (84)
Loss of appetite (Metabolism and nutrition disorders) | 21 (38)
Nausea (Gastrointestinal disorders) | 16 (37)
Diarrhea (Gastrointestinal disorders) | 17 (36)
Constipation (Gastrointestinal disorders) | 26 (86)
Sore throat (Gastrointestinal disorders) | 20 (38)
Stuffy nose (Respiratory, thoracic and mediastinal disorders) | 35 (85)
Fever (General disorders) | 16 (19)
Chills (General disorders) | 19 (32)
Rash (Skin and subcutaneous tissue disorders) | 13 (24)
Irritability (Psychiatric disorders) | 30 (76)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (2):
  • Informed Consent Form (2018-02-05): https://cdn.clinicaltrials.gov/large-docs/48/NCT02468648/ICF_000.pdf
  • Study Protocol and Statistical Analysis Plan (2019-11-25): https://cdn.clinicaltrials.gov/large-docs/48/NCT02468648/Prot_SAP_001.pdf